CLINICAL TRIAL: NCT04035187
Title: Prediction of Itraconazole Oral Absorption From In Vitro Dissolution
Brief Title: Itraconazole Oral Absorption
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, James E Polli, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00084585
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sequence A (fast, medium, oral solution, then slow) (Experimental): Participants first receive fast tablet, then medium tablet, then oral solution, and then slow tablet. Washout period is (at least) one week.
  Interventions: Drug: fast itraconazole tablet; Drug: medium itraconazole tablet; Drug: slow itraconazole tablet; Drug: oral itraconazole solution
- Sequence B (medium, slow, fast, then oral solution) (Experimental): Participants first receive medium tablet, then slow tablet, then fast tablet, and then oral solution. Washout period is (at least) one week.
  Interventions: Drug: fast itraconazole tablet; Drug: medium itraconazole tablet; Drug: slow itraconazole tablet; Drug: oral itraconazole solution
- Sequence C (slow, oral solution, medium, then fast) (Experimental): 3, 4, 2, 1 Participants first receive slow tablet, then oral solution, then medium tablet, then fast tablet. Washout period is (at least) one week.
  Interventions: Drug: fast itraconazole tablet; Drug: medium itraconazole tablet; Drug: slow itraconazole tablet; Drug: oral itraconazole solution
- Sequence D (oral solution, fast, slow, then medium) (Experimental): Participants first receive oral solution, fast tablet, then slow tablet, and then medium tablet. Washout period is (at least) one week.
  Interventions: Drug: fast itraconazole tablet; Drug: medium itraconazole tablet; Drug: slow itraconazole tablet; Drug: oral itraconazole solution

INTERVENTIONS:
Drug: fast itraconazole tablet — 100mg dose
  Other Names: fast dissolving itraconazole tablet
Drug: medium itraconazole tablet — 100mg dose
  Other Names: medium dissolving itraconazole tablet
Drug: slow itraconazole tablet — 100mg dose
  Other Names: slow dissolving itraconazole tablet
Drug: oral itraconazole solution — 100mg dose
  Other Names: commercial oral itraconazole solution

SUMMARY:
For tablets to be absorbed, the drug must dissolve after being swallowed. Drugs with low solubility sometimes require the inert ingredients in tablets to help the drug dissolve after being swallowed. This study uses itraconazole as an example drug with low solubility. Itraconazole tablets with different inert ingredients and manufacturing will be administered to healthy volunteers to see if the different inert ingredients and manufacturing impact drug absorption.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy, as determined by screening evaluation that is not greater than 30 days before the first drug study visit
* Subject is male or female between 18 and 65 years of age inclusive.
* Subject is an acceptable candidate for venipuncture.
* Subject is willing to stop all non-routine OTC medications, as well as vitamins, dietary supplements, and herbals, for 24 hours prior to study drug administration and during pharmacokinetic study visits.
* Subject is willing, for each of the four drug study periods, to stop consuming grapefruit, grapefruit products, star fruit, star fruit products, Seville oranges, and St. John's wort from 72-hour before study drug administration until the period's last blood sample
* Subject is willing to not smoke (or use e-cigarettes) during study visits.

Exclusion Criteria:

* Subject has a significant medical disease (including cardiovascular, pulmonary, hematologic, endocrine, immunologic, neurologic, gastrointestinal or psychiatric).
* Subject shows evidence of congestive heart failure or history of congestive heart failure.
* Subject exhibits electrocardiogram (12 lead) with clinically significant abnormalities (e.g. QTcF >450 msec).
* Subject has a history of alcohol or drug abuse, which in the opinion of the investigator, could jeopardize the subject's health or would compromise the subject's ability to participate in this trial.
* Subject is pregnant, breast feeding, or trying to become pregnant.
* Female subject of childbearing potential is unwilling or unable to use a medically acceptable method of contraception throughout the entire study period and for one week after the study is completed. Medically acceptable methods of contraception that may be used by the subject and/or her partner are: oral birth control pill, condom with spermicide, diaphragm with spermicide, IUD, vaginal spermicidal suppository, surgical sterilization of patient or their partner(s), abstinence, or hormonal-based patches, ring, injections, and implants.
* Subject routinely uses (i.e. daily or weekly) prescription medication except hormonal birth control medication, routinely uses (i.e. daily or weekly) OTC medication, or routinely uses (i.e. daily or weekly) St. John's Wort. OTC medications do not include vitamins, dietary supplements, or herbals.
* Subject routinely uses (i.e. daily or weekly) acid blockers, antacids, anti-diarrhea, stimulants, appetite suppressants, or anti-nausea medication or other drugs that modulate GI functio
* Subject is currently taking itraconazole or medication known to interact with itraconazole.
* Subject is allergic to itraconazole.
* Subject has liver impairment as assessed by alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin levels greater than the upper limit of normal (ULN).
* Subject has renal impairment as assessed by creatinine clearance lower than 50mL/min/1.73m2, using the CKD-EPI formula.
* Subject is not willing or able to be adherent to study protocol (e.g. study visits).
* Subject has a condition in which in the opinion of the PI or medical physician would increase risk to the subject or interfere with the integrity of the study.
* Subject has received an investigational product within 30 days prior to study drug administration, plans to receive an investigational product during their study participation period, or plans to donate blood to any other clinical trial during their study participation period.
* Subject has provided plasma donation within 1 month of screening or any blood donation/loss more than 500 mL within 8 weeks prior to study drug administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-05-21 (Actual); Study Completion 2022-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done through flyers and A/V advertisement throughout the University of Maryland Baltimore campus. Additionally, ResearchMatch.org was used. Planned initial interactions were phone calls and emails from potential subjects. Additionally, individuals who previously indicated a willingness to be contacted for future studies were contacted. Recruitment period was from September 17th 2019 to June 24th 2021.
Pre-assignment Details: Enrollment number is the number of participants who signed a consent form and passed screening tests.
Groups:
- Sequence C (Slow, Oral Solution, Medium, Then Fast): Participants first receive slow tablet, then oral solution, then medium tablet, then fast tablet. Washout period is (at least) one week.
  fast itraconazole tablet: 100mg dose
  medium itraconazole tablet: 100mg dose
  slow itraconazole tablet: 100mg dose
  oral itraconazole solution: 100mg dose
Period: Overall Study
Arm/Group | Sequence A (Fast, Medium, Oral Solution, Then Slow) | Sequence B (Medium, Slow, Fast, Then Oral Solution) | Sequence C (Slow, Oral Solution, Medium, Then Fast) | Sequence D (Oral Solution, Fast, Slow, Then Medium)
Started | 4 | 4 | 4 | 5
Completed | 2 | 2 | 4 | 4
Not Completed | 2 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0
Not completed — Participant lived out of state and due to COVID-19 pandemic could not travel to study site. | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A (Fast, Medium, Oral Solution, Then Slow) | Sequence B (Medium, Slow, Fast, Then Oral Solution) | Sequence C (Slow, Oral Solution, Medium, Then Fast) | Sequence D (Oral Solution, Fast, Slow, Then Medium) | Total
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 5 | 17
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (4.7) | 41.3 (12) | 28.3 (1.7) | 41 (15.3) | 34.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 2 | 10
  Male | 1 | 2 | 1 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 4 | 4 | 4 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 1 | 4
  White | 1 | 3 | 2 | 4 | 10
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: AUC
Description: area under the curve from 0-72hr
Time Frame: 0-72hr
Population: Seventeen participants were randomized in this cross-over study to receive all 4 itraconazole products at least one week apart. Twelve participants completed all 4 interventions. Analysis was only done of data from participants who completed all four interventions (n=12).
Measure: Mean (Standard Error); unit: ng*hr/mL
Groups:
- Fast Tablet: Fast-release itraconazole 100 mg tablet
- Medium Tablet: Medium-release itraconazole 100 mg tablet
- Slow Tablet: Slow-release itraconazole 100 mg tablet
- Oral Solution: Oral solution itraconazole 100 mg
Arm/Group | Fast Tablet | Medium Tablet | Slow Tablet | Oral Solution
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng*hr/mL | 1624.8 (146.1) | 1365.5 (184) | 1282.2 (220.3) | 1848.7 (139.7)

2. Secondary Outcome: Cmax
Description: maximum concentration during the time interval
Time Frame: 0-72hr
Population: Seventeen participants were randomized in this cross-over study to receive all 4 itraconazole products at least one week apart. Twelve participants completed all 4 interventions. Analysis was only done of data from participants who completed all four interventions.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Fast Tablet | Medium Tablet | Slow Tablet | Oral Solution
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng/mL | 174.3 (30.9) | 108.5 (14.9) | 121.3 (26.4) | 266.7 (40.5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time enrollment (signed consent) to the last study visit (72-hr blood draw time point).
Groups:
- Fast Tablet: All participants who received Fast-release itraconazole 100 mg tablet, regardless if they finish the cross-over study
- Medium Tablet: All participants who received Medium-release itraconazole 100 mg tablet, regardless if they finish the cross-over study
- Slow Tablet: All participants who received Slow-release itraconazole 100 mg tablet, regardless if they finish the cross-over study
- Oral Solution: All participants who received Oral solution itraconazole 100 mg tablet, regardless if they finish the cross-over study
Arm/Group | Fast Tablet | Medium Tablet | Slow Tablet | Oral Solution
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 3/14 | 1/14 | 1/13 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fast Tablet (N=14) | Medium Tablet (N=14) | Slow Tablet (N=13) | Oral Solution (N=12)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) — mild
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — mild
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — mild
Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT04035187/Prot_SAP_000.pdf